CLINICAL TRIAL: NCT01306799
Title: Effect of Chronic Proton Pump Inhibitor Therapy on Bone Mineral Density and Bone Structure in Mid to Late Adulthood
Brief Title: To Learn How Bone Structure and Bone Mass Change After Long-term PPI Use
Acronym: BE-CAST
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 810599; 1R01AR057102-01 (NIH)
Record Dates: First submitted 2011-02-17; First posted 2011-03-02 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Barrett's Esophagus; Erosive Esophagitis; Gastroesophageal Reflux Disease(GERD)
Keywords: Barrett's Esophagus; Erosive Esophagitis; Proton Pump Inhibitor (PPI); Bone; Bone Density; GERD; ulcer prophylaxis
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Barrett's Esophagus, Erosive Esophagitis, GERD

SUMMARY:
Patients with severe acid reflux and/or Barrett's esophagus are recommended to take Proton pump inhibitors (PPIs)indefinitely to prevent complications such as strictures or the development of a type of esophageal cancer. Recently, some studies suggested that taking these medications on a long-term basis may affect the bone. Therefore, it is important to learn whether these medications may lead to accelerated bone loss so that effective preventive measures can be developed for patients who require these medications for acid-related conditions. Several studies reported that patients receiving PPIs for many years may have increased risk of hip fractures. However, it is unclear whether this is because the PPIs cause reduced bone density or whether the increased risk of fractures has nothing to do with PPIs and is because patients who require PPIs have other illnesses that cause the increased fractures. The purpose of the study is to learn how bone structure and bone mass change after long-term PPI use.

DETAILED DESCRIPTION:
Proton pump inhibitors (PPIs) are among the most widely used medications. It is becoming increasingly common for patients to take these potent acid suppressants on a long-term and continuous basis for erosive esophagitis, Barrett's esophagus and protection against nonsteroidal anti-inflammatory drug-related gastropathy. PPI therapy leads to elevated serum gastrin levels and may impair the absorption of calcium and food-bound vitamin B12. PPI-induced hypergastrinemia has a direct trophic effect on the parathyroid glands, leading to parathyroid hyperplasia, increased parathyroid hormone secretion and bone loss. Furthermore, both calcium malabsorption and vitamin B12 deficiency are associated with reduced bone mineral density (BMD) and increased osteoporotic fracture risk. Consistent with these data, recent studies revealed a positive association between PPI therapy and the risk of osteoporotic fractures. Peripheral quantitative computed tomography (pQCT) can provide a three-dimensional structural analysis of trabecular and cortical volumetric BMD (vBMD) and dimensions. These data are imperative for a valid assessment of the effect of chronic PPI therapy on bone strength. The investigators hypothesize that PPI therapy leads to decreased cortical and trabecular vBMD, cortical dimensions and bone strength.

ELIGIBILITY:
Inclusion Criteria:

* women between 50 to 75 years old
* men between 40 to 75 years old
* Barrett's esophagus and Erosive esophagitis diagnosed within the past three years, GERD or Acid Reflux, taking chronic aspirin
* Starting long-term PPI therapy or currently on long-term PPI therapy

Exclusion Criteria:

* Pre-menopausal women
* men under 40 years old

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients who either are starting or have been receiving long-term continuous PPI therapy for erosive esophagitis or Barrett's esophagus diagnosed within the past three years.
  * Patients who are starting PPI therapy for gastroesophageal reflux disease (GERD) and have shown a subjective improvement in symptoms within 4 weeks of starting therapy. This improvement will be assessed either through documentation in their medical record or through telephone interview with permission from their physician.
  * Patients who are starting PPI therapy for ulcer prophylaxis in a setting of chronic aspirin use.
  * Patients who are starting PPI therapy for extraesophageal manifestations of GERD.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2010-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Volumetric bone mineral density as measured by pQCT | 3 years

SECONDARY OUTCOMES:
measure PTH levels at each study visit | 3 years
  monitor change in PTH levels because long-term PPI therapy may have an affect on parathyroid glands, increasing parathyroid hormone (PTH) secretion.
measure vitamin B12 levels at each study visit | 3 years
  low B12 levels have been associated with reduced bone mineral density (BMD) as well osteoporotic fracture risk

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Xiao Yang, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States